CLINICAL TRIAL: NCT01071291
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Period Crossover Study to Evaluate the Effects of Niaspan™ on Reverse Cholesterol Transport in Healthy Male Subjects
Brief Title: Effects of Niaspan™ on High-density Lipoprotein (HDL) in Healthy Male Subjects (0000-069)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-069; 069; 2010_510
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Arm A will receive a Niaspan treatment in Period 1 and Placebo treatment in Period 2
  Interventions: Drug: Niaspan; Drug: Comparator: Placebo
- Arm B (Experimental): Arm B will receive a Placebo treatment in Period 1 and Niaspan treatment in Period 2
  Interventions: Drug: Niaspan; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Niaspan — Niaspan™
  Other Names: NIASPAN™
Drug: Comparator: Placebo — Placebo

SUMMARY:
This study will evaluate whether chronic dosing with Niaspan™ increases reverse cholesterol transport, high-density lipoprotein cholesterol (HDL-C) levels, and fecal excretion of cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Subjects

Exclusion Criteria :

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cholesterol efflux | Baseline and 12 weeks
Change from the baseline in High-Density Lipoprotein Cholesterol (HDL-C) | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC